CLINICAL TRIAL: NCT00761826
Title: A Prospective Multicenter Trial To Evaluate The Safety And Effectiveness Of The MEL 80 Excimer Laser Using LASIK (Laser In Situ Keratomileusis) For The Correction Of Naturally Occuring Mixed Astigmatism Up To 6.0 D
Brief Title: Study of the MEL 80 Excimer Laser Using LASIK in the Treatment of Mixed Astigmatism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carl Zeiss Meditec, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEL 80-2006-2
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-01

CONDITIONS: Mixed Astigmatism
Keywords: Mixed Astigmatism; Laser In Situ Keratomileusis; Laser Therapy; Laser Corneal Surgery; Refractive Surgical Procedures; Ophthalmologic Surgical Procedure; Operative Surgical Procedures; Therapeutics
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: MEL 80 Mixed Astigmatism Treatment — Treatment of Naturally Occuring Mixed Astigmatic corrections up to 6.0 D.

SUMMARY:
The purpose of this study is to determine whether the MEL 80 Excimer Laser is effective in the treatment of mixed astigmatism up to 6.0 D, when used as part of the Laser In Situ Keratomileusis (LASIK) procedure.

DETAILED DESCRIPTION:
LASIK has become one of the most common refractive eye procedures performed in the country. In the mixed astigmatism procedure, a combination of both a steepening (hyperopic treatment) and a flattening (myopic treatment) occur on the corneal surface. The surgeon will produce a standard keratomileusis flap using a microkeratome, exposing the corneal stroma. Recontouring under the flap is then accomplished by the removal of tissue from the stroma with the laser. This recontouring results in an altering of effective lens power of the central cornea, measured in diopters (D). The MEL 80 Excimer Laser System will be evaluated for its ability to create accurate and stable mixed astigmatic refractive correction results.

ELIGIBILITY:
Inclusion Criteria:

* Naturally occurring mixed astigmatism when the magnitude of cylinder (up to 6.0 D) is greater than the magnitude of sphere, and the cylinder and sphere have opposite signs, at the spectacle plane;
* Have a stable refraction for at least the past twelve months, as demonstrated by a change of less than or equal to 0.50 D preoperative spherical equivalent shift over twelve months prior to surgery;
* Discontinue use of contact lenses at least 2 weeks for hard contacts and 3 days for soft lenses prior to the preoperative examination;
* Hard contact lens wearers must have two central keratometry readings and two manifest refractions taken at least one week apart that do not differ by more than 0.50 D
* Have visual acuity correctable to at least 20/40 in both eyes
* Have no more than 0.75 D of latent hyperopia as determined by the difference between the preoperative manifest refractive spherical equivalent (MRSE) and cycloplegic refractive spherical equivalent (CRSE);
* Be at least 18 years of age
* Corneal topography should be normal;
* The operative eye must be targeted for emmetropia;
* Be willing and able to return for scheduled follow-up examinations for twelve months after surgery;
* and provide written informed consent.

Exclusion Criteria:

* History of anterior segment pathology, including cataracts (in the operative eye);
* Clinically significant dry eye syndrome unresolved by treatment;
* Residual, recurrent, active ocular or uncontrolled eyelid disease, corneal scars within the ablation zone or other corneal abnormality such as recurrent corneal erosion or severe basement membrane disease;
* Ophthalmoscopic signs of keratoconus (or keratoconus suspect);
* Required ablation is deeper than 250 microns from the corneal endothelium;
* Irregular or unstable (distorted/not clear) corneal mires on central keratometry readings;
* Blind in the fellow eye;
* Previous intraocular or corneal surgery of any kind in the operative eye(s), including any type of surgery for either refractive or therapeutic purposes;
* History of ocular Herpes zoster or Herpes simplex keratitis;
* History of steroid-responsive rise in intraocular pressure, glaucoma, or preoperative IOP >21 mm Hg;
* Diabetes, diagnosed autoimmune disease, connective tissue disease or clinically significant atopic syndrome;
* Immunocompromised patients, or use of chronic systemic corticosteroid or other immunosuppressive therapy;
* Pregnant, lactating, or child-bearing potential and not practicing a medically approved method of birth control;
* Sensitivity to planned study medications;
* Simultaneous participation in other ophthalmic drug or device clinical trial.
* For Fellow (Second) Eyes in Simultaneous Bilateral Treatment Procedures
* 1. Flap complications during the first eye's surgery such as a free cap, partial flap, thin flap, or irregular flap.
* 2. Epithelial defect exceeding 2 mm x 2 mm in dimension, or clinically significant debris in the interface between the flap and underlying stroma for the first eye.
* 3. Severe blepharospasm in the first eye that may have prevented or impeded the completion of the keratectomy and/or the laser ablation procedure.
* 4. Poor subject cooperation with instructions for the first eye's surgery and/or poor subject fixation on the laser fixation target.
* 5. Aborted LASIK procedure in the first eye or PRK was performed in the first eye because LASIK was not possible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2007-01; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
At the point of stability, a minimum of 75% of eyes should have an achieved refraction within ± 1.00 D of the intended outcome, and at least 50% of eyes should be within ± 0.50 D of the intended outcome. | Point of stability
A minimum of 85% of eyes should have an uncorrected visual acuity of 20/40 or better at the postoperative interval at which stability has been established. | Point of stability
A minimum of 95% of eyes should have a change of < 1.00 D in manifest refraction spherical equivalent (MRSE) between 2 refractions performed at least 3 months apart, and the mean rate of MRSE change per month should be < 0.04 D. | Point of stability
Distance BSCVA of worse than 20/40 at the postoperative interval at which stability has been established should occur in less than 1.0 % of eyes that had a BSCVA of 20/20 or better before surgery. | Point of stability
Loss of more than 2 lines of BSCVA should occur in less than 5.0 % of eyes. | Postoperative visits
Incidence of adverse events to occur in less than 1% of eyes | Postoperative visits

SECONDARY OUTCOMES:
Subject Satisfaction: As measured by a subjective questionnaire, and will be considered as a secondary efficacy variable. | Postoperative visits 3, 6, 9 and 12 months
Incidence of complications | Postoperative visits
Patient Symptoms: As measured by a subjective questionnaire, will be considered as a secondary safety variable. | Preoperative and Postoperative visits 3, 6, 9 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: John Doane, MD, Principal Investigator — Discover Vision Centers; Richard Hoffman, MD, Principal Investigator — Fine, Hoffman, and Packer LLC; Howard Fine, MD, Principal Investigator — Fine, Hoffman, and Packer LLC; Mark Packer, MD, Principal Investigator — FIne, Hoffman, and Packer LLC; David Tanzer, MD, Principal Investigator — US Navy Refractive Surgery Center, San Diego, CA; John Vukich, MD, Principal Investigator — Davis Duehr Dean Eye Clinic; Jon Dishler, MD, Principal Investigator — Dishler Laser Institute
Locations (5):
- United States (5):
  - US Navy Refractive Surgery Center, San Diego, California
  - Dishler Laser Institute, Greenwood Village, Colorado
  - Discover Vision Centers, Kansas City, Missouri
  - Fine, Hoffman, and Packer, Eugene, Oregon
  - Davis Duehr Dean Eye Clinic, Madison, Wisconsin